CLINICAL TRIAL: NCT07102004
Title: A Phase I/II Study of MHB088C for Patients With Advanced Malignant Solid Tumors
Brief Title: Study of MHB088C for Patients With Advanced Solid Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHB088C-CP001CN
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Advanced/Metastatic Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MHB088C administered (Experimental): If needed, additional descriptive information (including which interventions are administered in each arm) to differentiate each arm from other arms in the clinical trial.
  Phase Ia:
  Participants with advanced solid tumor.
  Phase Ib:
  Participants with advanced solid tumor
  Phase II:
  Participants with advanced SCLC
  Interventions: Drug: MHB088C for Injection

INTERVENTIONS:
Drug: MHB088C for Injection — MHB088C for Injection, an antibody drug-conjugated molecule (ADC) MHB088C will be administered intravenously at a frequency of once every 2 weeks (Q2W) or every 3 week (Q3W).

SUMMARY:
This is a Phase I/II, multicenter, open-label clinical trial with dose escalation/dose expansion/efficacy expansion phases, designed to evaluate the safety/tolerability, pharmacokinetics, immunogenicity and preliminary efficacy of MHB088C in participants with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Agree to follow the experimental treatment plan and visit plan, join the group voluntarily, and sign a written informed consent form;
* Age ≥ 18 years old when signing the informed consent form;
* The Eastern Cooperative Oncology Group's physical status scoring standard (ECOG) is 0~1;
* The expected survival time is at least 3 months;
* Eligible participants of childbearing potential must agree to take highly reliable contraceptive measures with their partners during the study and within at least 90 days after the last dose and agree not to retrieve, freeze or donate sperm or ova from screening to at least 3 months after the last dose of investigational drug; female participants of childbearing potential must have a negative results of blood pregnancy test before the first dose of investigational drug, and must be non-lactating.
* Understand study requirements, willing and able to comply with study and follow-up procedures.

Neoplasm-related criteria

* Phase Ia: Histologically or cytologically confirmed unresectable advanced or metastatic malignant solid tumors, that is progressed or intolerant with standard of care (SOC), or for which no SOC regimens are available.
* Phase Ib: Histologically or cytologically confirmed unresectable advanced or metastatic malignant solid tumors, that is relapsed or progressed following systemic treatment or no SOC is available;
* Phase II: Histologically or cytologically documented unresectable advanced or metastatic SCLC and previous progressed during or after platinum-contained chemotherapy and immune-checkpoint inhibitors (ICIs).

Exclusion Criteria:

* Has more than 2 primary malignancies before signing of Informed Consent Form.
* Has received anti-tumor treatment before the first dose of investigational product; Medication of traditional Chinese medicine before the first dose of investigational drug.
* Medication of other unmarketed investigational drugs or therapies before the first dose of investigational drug.
* Presence of unstable brain metastases and/or leptomeningeal carcinomatosis.
* Has adverse reactions from previous anti-tumor treatment that have not recovered to ≤ CTCAE 5.0 Grade 1;
* Has underwent major organ surgery or significant trauma before the first dose of investigational drug or requiring elective surgery during the study.
* Has vaccinated with attenuated live vaccines before the first dose of investigational drug.
* Has mucosal or internal bleeding for non-traumatic reason before the first dose of investigational drug.
* Has received treatment with systemic corticosteroids or other immunosuppressive agents before the first dose of investigational drug.
* Has pulmonary disease that severely impact pulmonary function.
* Has history of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, or current ILD/pneumonia, or suspected ILD/pneumonia that cannot be excluded by imaging examination at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Adverse event (AE) and Serious adverse event (SAE) (Phase Ia) | After first administration of study drug until 30 days after last dose of study drug. Through phase Ia completion, an average of 1 year.
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)
Dose limited toxicity (DLT) (Phase Ia) | Cycle 1 (28 days for subjects receiving a dosing frequency of every 2 weeks, or 21 days for subjects receiving a dosing frequency of every 3 weeks)
  The DLTs of MHB088C will be determined.
Maximum tolerated dose (MTD) (Phase Ia) | Cycle 1 (28 days for subjects receiving a dosing frequency of every 2 weeks, or 21 days for subjects receiving a dosing frequency of every 3 weeks).
  The maximum tolerated dose (MTD) of MHB088C will be evaluated on the first cycle.
Recommended phase II dose (RP2D) (Phase Ib) | Through phase Ib completion, an average of 1 year.
  RP2D will be selected upon safety, PK and efficacy data.
Objective response rate (ORR) (phase II) | Approximately 48 months.
  The ORR is defined as the proportion of subjects with confirmed complete response (CR) or confirmed partial response (PR), based on RECIST Version 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China